CLINICAL TRIAL: NCT00376714
Title: A Randomised, Double-Blind, Placebo-Controlled, Dose Ascending, 3 Period Crossover Study To Examine The Safety, Tolerability, Pharmacodynamics And Pharmacokinetics Of Repeat Inhaled Doses Of GSK233705B In COPD Subjects.
Brief Title: Safety And Tolerability Study In Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: AC2105333
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: plethysmography; muscarinic receptor antagonist; COPD; repeat dosing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK233705

SUMMARY:
GSK233705 is a high-affinity specific muscarinic receptor (mAChR) antagonist which is being developed for once daily treatment of chronic obstructive pulmonary disease (COPD). The long duration of action of GSK233705 when administered via inhalation in animal models supports the potential for use as a once-daily bronchodilator for chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be of non-childbearing potential including pre-menopausal females
* Male subjects must agree to abstain from or use a condom during sexual intercourse with pregnant or lactating females
* Subject diagnosed with COPD, as defined by the GOLD guidelines
* Body weight greater than 50kg
* Subject is a smoker or an ex-smoker with a smoking history of at least 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or equivalent).
* Subject has FEV1/FVC < 0.7 post-bronchodilator (salbutamol).
* Subject has FEV1 greater than or equal to 80% of predicted normal for height, age and gender after inhalation of 200 µg salbutamol.
* Response to ipratropium bromide defined as:
* Either: An increase in FEV1 of =12% and =150 mL at 2 h following inhalation of 80 ug of ipratropium bromide at the screening visit
* or: a documented increase in FEV1 of =12% and =150 mL at 2 h following inhalation of 80 ug of ipratropium bromide within 6 months of screening and an increase in FEV1 of >6% and >100ml 2h following inhalation of 80 ug of ipratropium bromide at the screening visit (in order to allow for potential fluctuations in the response to ipratropium bromide in patients known to be responders to ipratropium bromide).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subject is available to complete all study measurements and procedures.

Exclusion Criteria:

* Subjects who have a past or present disease, judged by the Investigator and the Medical Monitor, to affect the outcome of this study.
* The subject has a positive urine drug/ urine alcohol screen.
* History of alcohol/drug abuse or dependence within 12 months of the study:
* The subject has a positive pregnancy test.
* Subject has FEV1 greater than or equal to 40% of predicted after inhalation of salbutamol.
* A positive Hepatitis B or Hepatitis C result within 3 months of screening
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period
* The subject has donated a unit of blood within 30 days of screening, or, intends to donate during the study.
* Subject has claustrophobia that may be aggravated by entering the plethysmography cabinet.
* The subject has a known allergy or hypersensitivity to ipratropium bromide, tiotropium bromide, atropine and any of its derivatives or milk protein/lactose.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* Subject is unable to use the DISKUS™ device correctly.
* Subject has prostate hypertrophy or narrow angle glaucoma.
* Use of prescription drugs (with the exception of those allowed in the protocol) and herbal remedies (e.g. St John's Wort) within 48 hours of each treatment period

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2006-08-16; Study Completion 2007-04-03 (Actual)

PRIMARY OUTCOMES:
Adverse events Blood pressure Heart rate 12-lead ECG Holter monitoring Lead II ECG monitoring Lung function Clinical laboratory safety tests.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) Serial specific airways conductance (sGaw), airways resistance (Raw) Rescue medication usage Plasma and urine concentrations of GSK233705 and derived pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: AC2105333 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AC2105333 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC2105333 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AC2105333 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC2105333 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC2105333 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AC2105333 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register